CLINICAL TRIAL: NCT02026505
Title: Prospective Assessment of the Cardiac Effects the Proteasome Inhibitor Bortezomib in Patients Undergoing Therapy for Multiple Myeloma
Brief Title: Evaluation of Cardiotoxic Effects of Bortezomib
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: Millennium: The Takeda Oncology Company (Industry)
Responsible Party: Principal Investigator, Stephen Heitner, Assistant Professor of Medicine, Oregon Health and Science University
Other Study IDs: IRB00010254
Record Dates: First submitted 2013-12-18; First posted 2014-01-03 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Multiple Myeloma; Heart Failure, Systolic; Cardiotoxins
MeSH Terms: conditions — Multiple Myeloma; Heart Failure, Systolic | interventions — Bortezomib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood and serum for batch analysis. Once the assays have been completed, the samples will be discarded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple Myeloma, Bortezomib
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib

SUMMARY:
The purpose of this study is to learn more about how a drug commonly used to treat multiple myeloma can affect the heart.

In this study, the investigators will learn whether a drug called how a drug (called bortezomib, or Velcade) receive for multiple myeloma affects the heart. Bortezomib is part of the standard treatment and its effects on multiple myeloma is not being studied here.

The investigators want to learn whether damage occurs to the heart after taking bortezomib for multiple myeloma, whether it is reversible, and we can predict damage to the heart before it occurs.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of multiple myeloma
* have a treatment plan involving greater than 4 cycles of bortezomib-based chemotherapy

Exclusion Criteria:

* pre-existing history of left ventricular systolic dysfunction
* congestive heart failure
* coronary artery disease
* significant valvular heart disease
* cardiac arrhythmias
* estimated glomerular filtration rate <30 mL/min/1.73m2

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (>18 years and <70 years) with multiple myeloma
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Global longitudinal strain by echocardiography | 6 months

SECONDARY OUTCOMES:
Amount of late gadolinium enhancement by cardiac MRI | 6 months
High-sensitivity troponin T | 6 months
C-reactive protein | 6 months
Serum NT-proBNP | 6 months
Carboxyl-terminal telopeptide of collagen type I | 6 months
Amino-terminal peptide of procollagen type III | 6 months